CLINICAL TRIAL: NCT00705887
Title: The Feasibility of a Motivational Enhancement Approach to Skin Cancer Prevention in a Sample of Young Adult Patients
Brief Title: A Motivational Enhancement Approach to Skin Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Christina P. Linton, FNP-BC, PhD, Oregon Health & Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00002996
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-06

CONDITIONS: Ultraviolet Rays; Motivation
Keywords: Ultraviolet Rays; Motivation; Health Education; Randomized Controlled Trial; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Health Education; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Brochure from the American Academy of Dermatology on protecting your skin from UV rays.
- Intervention (Experimental): Participation in a brief motivational enhancement session. These participants also received the same American Academy of Dermatology brochure on protecting your skin from UV rays.
  Interventions: Behavioral: Brief Motivational Enhancement Intervention

INTERVENTIONS:
Behavioral: Brief Motivational Enhancement Intervention — The motivational enhancement intervention lasted 5-8 minutes and consisted of gaining the client's permission to address the topic of skin cancer prevention, exchanging information through the elicit-provide-elicit strategy of information exchange, and summarization/ conclusion based on verbal and nonverbal cues from the participant.
  Other Names: Adaptation of Motivational Interviewing
  Arms: Intervention

SUMMARY:
The specific aims of this research are:

Aim 1 - To describe the UV protection behaviors and beliefs of young adult patients in a dermatology clinic.

Aim 2 - To examine whether or not the UV protection behaviors and beliefs of young adult dermatology patients are associated with age, gender, level of education, marital status, contact with skin cancer, time outdoors, skin type, the reason for their visit, and the date of data collection.

Aim 3 - To test the efficacy of a motivational enhancement approach to UV protection counseling for young adult dermatology patients, as manifested by favorable changes in UV protection stages of change, UV protection self-efficacy, and UV protection attitudes.

DETAILED DESCRIPTION:
Although skin cancer is the most common form of cancer in the United States, it is highly preventable by reducing exposure to ultraviolet (UV) radiation. However, recent primary prevention efforts have been inadequate in evoking behavior change, as manifested by increasing rates of ultraviolet radiation exposure, particularly among young adults. These findings indicate the need to research novel approaches to skin cancer prevention.

Motivational enhancement techniques facilitate patient-centered, directive discussions wherein practitioners provide clear structure and encourage patients to play an active role in the consultation. The use of motivational enhancement techniques for health behavior change in medical settings has thus far yielded encouraging results for other health behavior change topics, but research has not yet investigated the application of these techniques to skin cancer prevention discussions.

ELIGIBILITY:
Inclusion Criteria:

* Dermatology patient presenting for scheduled appointment
* 18-30 years old

Exclusion Criteria:

* Seeking treatment for sunburn
* Unable to read and understand English
* Having previously received medical treatment from the interventionist

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
UV Protection Stages of Change | 6 months

SECONDARY OUTCOMES:
UV Protection Attitudes | 6 months
UV Protection Self-Efficacy | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Christina P Linton, FNP-BC, PhD, Principal Investigator — Oregon Health and Science University; Nancy Press, PhD, Study Chair — Oregon Health and Science University
Locations (1):
- Central Utah Clinic, Dermatology, Provo, Utah, United States